CLINICAL TRIAL: NCT04325373
Title: Study of Thrombotic Complications After Abdominal Aortic Aneurysm Surgery With or Without Infection: AAA-IT
Brief Title: Abdominal Aortic Aneurysm Surgery and Thrombosis
Acronym: AAA-IT
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2020/07
Record Dates: First submitted 2020-03-09; First posted 2020-03-27 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: abdominal aortic aneurysm; NETosis; thrombosis
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of our study is to evaluate the incidence of post-operative thrombotic complications after abdominal aortic aneurysm surgery in the context of atherosclerosis or infectious aneurysm and its links with preoperative inflammation and hemostasis.

DETAILED DESCRIPTION:
Abdominal aortic aneurysm (AAA) develops in the context of atherosclerosis or infection (aortitis or mycotic aneurysm). AAA and its surgery are associated with pro-thrombotic modifications of hemostasis, which persists in the post-operative period. Pro-thrombotic reactions occur in the intraluminal thrombus. Inflammatory cells recruitment is mediated by adhesion molecules from the activated endothelium, such as "vascular cell adhesion molecule-1" (VCAM-1), "intercellular adhesion molecule-1" (ICAM-1), P-selectin and E-selectin.

In the setting of infection, neutrophil death process occurs, the NETosis, with the liberation of Neutrophil Extracellular Traps (NETs), containing DNA and histones. NETs are associated with thrombosis and various studies have already quantified NETosis biomarkers in plasma from patients with thrombotic disease, such as MPO-DNA (DNA coupled myeloperoxidase).

In the clinical perioperative setting, patients with aortitis scheduled for AAA surgery shwoed exhibit thrombotic events.

The hypothesize was that patients with aortitis have an inflammatory and hemostatic activation different from patients who develop AAA in atherosclerotic condition, and that inflammation is a risk factor of postoperative thrombotic events.

ELIGIBILITY:
Inclusion Criteria:

* patient >18 years-old;
* patient scheduled for AAA surgery by laparotomy in the vascular surgical unit at Bordeaux University Hospital;
* patient who gave his/her authorization for the use of its medical data and results of blood analyses performed on residual plasma and results of aortic material analyses

Exclusion Criteria:

* patient who do not understand the study (not fluently French speaking or unable to give his/her consent);
* patient with a pre-existing hemostatic disorder;
* patient scheduled for an endovascular surgery and benefiting from a secondary laparotomy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with surgery for abdominal aortic aneurysm
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2021-01-27 (Actual); Study Completion 2021-01-27 (Actual)

PRIMARY OUTCOMES:
thrombotic events | first 7 postoperative days after AAA surgery
  Incidence of thrombotic events

SECONDARY OUTCOMES:
white blood cells | baseline
  white blood cells (G/L),
hemoglobin | baseline
  hemoglobin (g/dL),
platelets | baseline
  platelets (G/L),
prothrombin time ratio | baseline
  prothrombin time ratio (%),
INR | baseline
  INR
aPTT ratio | baseline
  aPTT ratio
fibrinogen | baseline
  fibrinogen (g/L),
CRP | baseline
  CRP (ng/mL),
interleukin-6 | baseline
  interleukin-6 (pg/mL),
thrombin generation test | baseline
  thrombin generation test (lag time (min),
peak | baseline
  peak (nM),
time to peak | baseline
  time to peak (min),
ETP | baseline
  ETP (nM.min),
velocity index | baseline
  velocity index
von Willebrand factor | baseline
  von Willebrand factor (%),
soluble P-selectin | baseline
  soluble P-selectin (ng/mL),
MPO-AND | baseline
  MPO-AND (% standard)
atherosclerosis | baseline
  % of patients with preoperative atherosclerosis (number)
Aspirin treatment | baseline
  % of patients with preoperative treatment by Aspirin (number)
clamping duration | baseline
  clamping duration (min),
bleeding | baseline
  bleeding (min),
vascular filling | baseline
  vascular filling (ml),
tranexamic acid administration | baseline
  tranexamic acid administration (g),
transfusion | baseline
  transfusion (pack of red blood cells, plasma volume (ml),
amount of fibrinogen | baseline
  amount of fibrinogen (g),
amount of heparin | baseline
  amount of heparin (UI)
Type of postoperative anticoagulation | baseline
  Type of postoperative anticoagulation: % of patients with unfractionated heparin or low-molecular-weight heparin
Administration way of postoperative anticoagulation | Baseline
  Administration way of postoperative anticoagulation: % of administration intra-venous or subcutaneously

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No